CLINICAL TRIAL: NCT00593645
Title: A Non-Myeloablative Conditioning Regimen for Allogeneic Transplantation With Clofarabine, Cytarabine, and Thymoglobulin for Myelodysplastic Syndrome and Acute Myeloid Leukemia
Brief Title: Clofarabine, Cytarabine, and Thymoglobulin for Allogeneic Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: toxicities were worse than expected
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-0702; No grant number
Record Dates: First submitted 2008-01-02; First posted 2008-01-15 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia
Keywords: Conditioning regimens; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Allogeneic Stem Cell Transplantation; Nonmyeloablative conditioning; Clofarabine; Cytarabine; Anti-thymocyte globulin
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Clofarabine; Cytarabine; thymoglobulin; Antilymphocyte Serum; Stem Cell Transplantation; Peripheral Blood Stem Cell Transplantation; Bone Marrow Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1: Non-myeloablative conditioning regimen (Experimental): * Clofarabine 40mg/m2/day IV over two hours daily x 5 days on Days -6 thru -2
  * Cytarabine 1gm/m2/day IV over two hours daily x 5 days on Days -6 thru -2 after the START of Clofarabine.
  * Thymoglobulin 1.0mg/kg IV over 6 hours X 1 day on Day -4, then 2.5mg/kg/day x 2 days on Days -3 and -2.
  * Stem Cell Transplant - On day 0 a minimum of total CD34+ cell dose of 2 x10E6/kg (actual weight of recipient) will be infused.
  Interventions: Drug: Clofarabine; Drug: Cytarabine; Drug: Thymoglobulin; Procedure: Stem cell infusion

INTERVENTIONS:
Drug: Clofarabine
  Other Names: Clolar
Drug: Cytarabine
  Other Names: Ara-C; Cytosar
Drug: Thymoglobulin
  Other Names: Anti-thymocyte globulin
Procedure: Stem cell infusion
  Other Names: Stem cell transplant; Hematopoietic stem cell transplant; Peripheral blood stem cell transplant; Bone marrow transplant

SUMMARY:
This study will test the combination of clofarabine, cytarabine, and thymoglobulin as a non-myeloablative conditioning regimen for patients with myelodysplastic syndromes or acute myeloid leukemia undergoing allogeneic stem cell transplant.

DETAILED DESCRIPTION:
Current reduced intensity conditioning regimens have been able to decrease TRM (treatment related mortality) but suffer from increased rates of disease relapse. Disease burden at transplantation, as measured by percent myeloblasts, predicts relapse. Current regimens employ fludarabine and busulfan with various adjutants, but these agents are not part of the usual armamentarium used versus leukemia and have questionable anti-leukemic activity. By substituting clofarabine and cytarabine, a combination with proven anti-leukemic activity in the relapsed and refractory setting as well as activity versus MDS, as the back bone of the regimen we hope overcome residual disease and improve post-transplant relapse rates. Furthermore the principal toxicity of this regimen is myelosuppression, which should be abrogated by the infusion of stem cells. Thymoglobulin is included due to its minimal contribution to toxicity but significant benefits in engraftment, and controlling acute and chronic GVHD, which are major contributors to TRM and disease specific activity in MDS.

ELIGIBILITY:
Inclusion Criteria (Patient):

1. Myelodysplastic Syndrome (MDS), as defined by the World Health Organization criteria, OR Chronic Myelomonocytic Leukemia (CMML) as defined by the French American British classification OR Acute Myeloid Leukemia (AML) in complete remission [excluding FAB-M3] diagnosed by standard criteria and meet the criteria below:

   1. Patients may be in any CR
   2. No more than 2 cycles of consolidation. Any consolidation regimen may be used.
   3. No more than 6 months from documented CR to transplant.
2. Age 18 years or older.
3. ECOG performance status <=2
4. Identification of suitable donor
5. DLCO >=40% with no symptomatic pulmonary disease
6. LVEF by MUGA >= 30%
7. Serum creatinine <=1.0 mg/dL; if serum creatinine >1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be >60 mL/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease equation where Predicted GFR (ml/min/1.73 m2) = 186 x (Serum Creatinine)-1.154 x (age in years)-0.023 x (0.742 if patient is female) x (1.212 if patient is black).
8. Bilirubin <=2 times the upper limit of normal
9. AST <=3 times the upper limit of normal

Donor criteria:

1. HLA-Matched Sibling: The donor must be an adequate HLA match as determined by serologic typing for class (A, B) and low resolution molecular typing for class II (DRB1) as defined by institutional standards.
2. Matched Unrelated Donor: An acceptable match per NMDP standards based on high resolution molecular typing.
3. The donor must be healthy and must be an acceptable donor as per institutional standards for stem cell collection.
4. The donor must have no significant cardiopulmonary, renal, endocrine, or hepatic disease.
5. There is no upper age restriction for donors, but they must be at least 18 years of age.
6. Syngeneic donors are not eligible.
7. No known HIV.

Exclusion Criteria:

1. Pregnant or nursing.
2. Active systemic infection considered opportunistic, life threatening or clinically significant at the time of treatment.
3. Severe concurrent disease, including severe insulin-dependent diabetes, uncontrolled hypertension, transient ischemic attacks, uncontrolled symptomatic coronary artery disease, or symptomatic CNS involvement or psychiatric illness/social situations that would limit compliance with study requirements.
4. Known HIV disease.
5. History of other malignancy except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast unless the subject has been off treatment and free from disease for > 3 years.
6. Active disease at the time of transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Vij, M.D., Principal Investigator — Washington Universtiy of St. Louis
Locations (1):
- Ravi Vij, M.D., St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment to the study opened on 11/21/2007 and enrollment to the study closed on 08/11/2008
Period: Overall Study
Arm/Group | Arm 1: Non-myeloablative Conditioning Regimen
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1: Non-myeloablative Conditioning Regimen
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 54 [24 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 7
Diagnosis [Number; unit: participants]
  Myelodysplastic syndrome | 3
  Acute myeloid leukemia | 4

OUTCOME MEASURES:

1. Primary Outcome: Six-month Treatment Related Mortality
Time Frame: 6 months
Population: This outcome was not analyzed.
  Enrollment to the trial was halted after three of the first seven patients expired. This fulfilled the predefined stopping rule as it was unlikely that we would achieve our primary end point of a 6 month treatment-related mortality of 10%.
Arm/Group | Arm 1: Non-myeloablative Conditioning Regimen
Number analyzed (Participants) | 0

2. Secondary Outcome: Disease Specific Response Rates
Description: Disease-specific partial response and complete response.
Time Frame: One, three, six and twelve months.
Population: This outcome was not analyzed due to terminating the study after 7 participants were enrolled.
  We felt that the engraftment as measured by percent donor chimerism provided better response details than the limited data that was collected for the disease specific partial and complete response rates.
Arm/Group | Arm 1: Non-myeloablative Conditioning Regimen
Number analyzed (Participants) | 0

3. Secondary Outcome: Engraftment as Measured by Percent Donor Chimerism
Time Frame: Day +30
Population: 2 participants were not analyzed because they expired prior to Day +30.
Measure: Number; unit: participants
Arm/Group | Arm 1: Non-myeloablative Conditioning Regimen
Number analyzed (Participants) | 5
participants
  Not done | 2
  50% donor (bone marrow) | 1
  100% donor (bone marrow) | 1
  23.5% donor (FISH) | 1

4. Secondary Outcome: Engraftment as Measured by Percent Donor Chimerism
Time Frame: Day +40-+60
Population: 3 participants were not analyzed because they were expired.
Measure: Number; unit: participants
Arm/Group | Arm 1: Non-myeloablative Conditioning Regimen
Number analyzed (Participants) | 4
participants
  60% donor (bone marrow) | 1
  70% donor (bone marrow) | 1
  75% donor (bone marrow) | 1
  100% donor (peripheral blood) | 1

5. Secondary Outcome: Engraftment as Measured by Percent Donor Chimerism
Time Frame: Day +80-+90
Population: 3 participants were not analyzed as they were deceased.
Measure: Number; unit: participants
Arm/Group | Arm 1: Non-myeloablative Conditioning Regimen
Number analyzed (Participants) | 4
participants
  0% donor | 1
  33% donor - myeloid (peripheral blood) | 1
  67% donor (bone marrow) | 1
  100% donor (bone marrow) | 1

6. Secondary Outcome: Overall Survival
Time Frame: 5 years from time of restaging
Measure: Median (Full Range); unit: days
Arm/Group | Arm 1: Non-myeloablative Conditioning Regimen
Number analyzed (Participants) | 7
days | 237 [15 to 443]

7. Secondary Outcome: Disease-free Survival
Description: Disease-free survival is defined as the length of time after treatment ends that the participant survives without any signs or symptoms of that cancer.
Time Frame: 5 years from time of restaging
Population: None of the patients analyzed survived without any signs or symptoms of that cancer.
Measure: Number; unit: participants
Arm/Group | Arm 1: Non-myeloablative Conditioning Regimen
Number analyzed (Participants) | 7
participants | 0

8. Secondary Outcome: Rate of Acute Graft-versus-host Disease (GVHD)
Description: Acute GVHD occurs within 100 days of transplant.
Time Frame: Up to 100 days after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Non-myeloablative Conditioning Regimen
Number analyzed (Participants) | 7
percentage of participants | 0

9. Secondary Outcome: Rate of Chronic Graft-versus-host Disease (GVHD)
Time Frame: 100 days-1 year after transplant
Population: None of the participants had chronic graft-versus-host disease (GVHD). 3 participants expired prior to day 100.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Non-myeloablative Conditioning Regimen
Number analyzed (Participants) | 4
percentage of participants | 0

10. Secondary Outcome: Use Conventional STR-PCR Method for Monitoring Engraftment
Description: Includes assessment of mixed chimerism in the whole blood, myeloid cells, T cells, and B cells.
Time Frame: Up to 1 year after transplant
Population: This outcome was not analyzed specifically as the conventional STR-PCR method was used for monitoring engraftment.
Arm/Group | Arm 1: Non-myeloablative Conditioning Regimen
Number analyzed (Participants) | 0

11. Secondary Outcome: Median Time to Progression
Description: Time to progression is defined as the length of time from the start of treatment until the disease starts to get worse or spread to other parts of the body.
Time Frame: 5 years from time of restaging
Population: Of the four surviving patients, three relapsed. One patient remained in remission on day +120.
Measure: Median (Full Range); unit: days
Arm/Group | Arm 1: Non-myeloablative Conditioning Regimen
Number analyzed (Participants) | 3
days | 152 [98 to 154]

ADVERSE EVENTS:
Time Frame: Adverse event collection started from the beginning of treatment through 1 year post transplant.
Groups:
- Arm 1: * Clofarabine 40mg/m2/day IV over two hours daily x 5 days on Days -6 thru -2
  * Cytarabine 1gm/m2/day IV over two hours daily x 5 days on Days -6 thru -2 after the START of Clofarabine.
  * Thymoglobulin 1.0mg/kg IV over 6 hours X 1 day on Day -4, then 2.5mg/kg/day x 2 days on Days -3 and -2.
  * Stem Cell Transplant - On day 0 a minimum of total CD34+ cell dose of 2 x10E6/kg (actual weight of recipient) will be infused.
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 5/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=7)
Bilirubin (Investigations) | 1
Chest pain (Cardiac disorders) | 1
Death - respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 — Patient died on day +26 of veno-occlusive disease
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Infection with Gr. 3/4 neutropenia (Infections and infestations) | 1 — Sepsis - Resulted in (2) deaths on day +15 and day +32
Mucositis (Gastrointestinal disorders) | 1
Perforation, GI - colon (Gastrointestinal disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Seizure (Nervous system disorders) | 1
Uric acid (Metabolism and nutrition disorders) | 1
Death due to disease progression (General disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=7)
Abdominal pain (Gastrointestinal disorders) | 3
Acute renal failure (Renal and urinary disorders) | 2
Alkaline phosphatase (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3
Atrial fibrillation (Cardiac disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Blood blister - chin (Skin and subcutaneous tissue disorders) | 1
Blurred vision (Eye disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 1
CNS hemorrhage (Nervous system disorders) | 1
Catheter site (Injury, poisoning and procedural complications) | 2
Chest pain (Cardiac disorders) | 4
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Cystitis (Renal and urinary disorders) | 4
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2
Dental: teeth (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 7
Distension/bloating (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysgeusia/taste alteration (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Edema - right eyelid (Eye disorders) | 1
Edema:limb (General disorders) | 7
Elevated creatinine (Investigations) | 4
Elevated uric acid (Investigations) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Extremity pain (Musculoskeletal and connective tissue disorders) | 7
Eye hemorrage (Eye disorders) | 2
Fatigue (General disorders) | 5
Fever in the absence of neutropenia (General disorders) | 3
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Generalized edema (General disorders) | 1
Generalized pain (General disorders) | 1
Generalized weakness (General disorders) | 5
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 4
Hard of hearing (Ear and labyrinth disorders) | 1
Headache (Nervous system disorders) | 3
Hemianopsia (Eye disorders) | 1
Hemoglobin (Investigations) | 3
Hemorrhoids (Gastrointestinal disorders) | 1
Hot flashes (Vascular disorders) | 1
Hyperbilirubinemia (Investigations) | 5
Hyperglycemia (Investigations) | 4
Hyperkalemia (Investigations) | 4
Hypermagnesemia (Investigations) | 1
Hypernatremia (Investigations) | 2
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Hypertension (Cardiac disorders) | 4
Hypoalbuminemia (Investigations) | 6
Hypocalcemia (Investigations) | 5
Hypoglycemia (Investigations) | 1
Hypokalemia (Investigations) | 6
Hypomagnesemia (Investigations) | 5
Hyponatremia (Investigations) | 3
Hypotension (Cardiac disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Infection with Gr. 3-4 neutrophils (Infections and infestations) | 5
Infection with normal neutrophils (Infections and infestations) | 3
Infectious colitis (Infections and infestations) | 1
Insomnia (Psychiatric disorders) | 2
Keratitis (Eye disorders) | 1
Leukocytes (WBC) (Investigations) | 5
Leukoplakia (Gastrointestinal disorders) | 1
Line erythema/ecchymosis (Skin and subcutaneous tissue disorders) | 3
Liver abscess (Infections and infestations) | 1
Lower gastrointestinal hemorrhage (NOS) (Gastrointestinal disorders) | 2
Lymphopenia (Investigations) | 5
Mental status change (Psychiatric disorders) | 1
Mucositis (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 5
Neck/chin pain (Musculoskeletal and connective tissue disorders) | 2
Neuropathy - sensory (Nervous system disorders) | 3
Neutropenic fever (Infections and infestations) | 7
Neutrophils (Investigations) | 5
Petechiae (Skin and subcutaneous tissue disorders) | 3
Platelets (Investigations) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Poor vision (Eye disorders) | 1
Pruritis/itching (Skin and subcutaneous tissue disorders) | 1
Ptosis (Nervous system disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6
Right-sided weakness (Musculoskeletal and connective tissue disorders) | 1
Rigors/chills (General disorders) | 6
SGOT (AST) (Investigations) | 7
SGPT (ALT) (Investigations) | 7
Scrotal chafing (Skin and subcutaneous tissue disorders) | 1
Sinus bradycardia (Cardiac disorders) | 2
Somnolence (Nervous system disorders) | 1
Tachycardia (Cardiac disorders) | 3
Urinary frequency/urgency (Renal and urinary disorders) | 2
Urinary hesitancy (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 6

LIMITATIONS AND CAVEATS:
Enrollment was halted after 3 of the first 7 patients expired on days 15/26/32. Predefined early stopping rules were defined that if three deaths occurred in the first 11 patients then it was unlikely to achieve a low treatment-related mortality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes